CLINICAL TRIAL: NCT00376623
Title: An Open, Randomised Clinical Phase II Trial to Investigate the Efficacy, Safety and Pharmacokinetics of a Single Dose of 200 mg of i.v. BI 2536 in Comparison to 50 mg of i.v. BI 2536 Administered on Days 1, 2 and 3 in Patients With Advanced or Metastatic Non Small Cell Lung Cancer
Brief Title: Efficacy and Safety of BI 2536 in Advanced or Metastatic Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1216.9
Record Dates: First submitted 2006-09-14; First posted 2006-09-15 (Estimated); Results first posted 2022-05-06 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — BI 2536

ARMS (3):
- 200 milligram (mg) of BI 2536 (Experimental): Day 1
  Interventions: Drug: BI 2536
- 50 milligram (mg) of BI 2536 (Experimental): Day 1, 2, and 3
  Interventions: Drug: BI 2536
- 60 milligram (mg) of BI 2536 (Experimental): Day 1, 2, and 3
  Interventions: Drug: BI 2536

INTERVENTIONS:
Drug: BI 2536 — Intravenous Infusion

SUMMARY:
The trial will be performed to evaluate whether BI 2536 may be effective in the treatment of advanced or metastatic NSCLC of stage IIIB or IV in patients who relapsed after or failed first-line therapy. A secondary aim is to identify the most suitable dosage schedule for the further Phase II and III clinical programme of BI 2536. To achieve this objective two dosage schedules are compared.

ELIGIBILITY:
Inclusion Criteria:

male or female patients aged 18 years or older with histologically or cytologically confirmed advanced or metastatic NSCLC of stage IIIB or IV, who relapsed or failed prior first-line chemotherapy for advanced or metastatic disease. At least one tumour lesion must be present that can accurately be measured by magnetic resonance imaging (MRI), or computed tomography (CT) in at least one dimension (longest diameter to be recorded) as 20 mm or greater with conventional techniques or as 10 mm or greater with spiral CT scan. Life expectancy of at least three months; Eastern co-operative oncology group (ECOG) performance score of 2 or less and written informed consent which must be consistent with international conference on harmonisation good clinical practice (ICH-GCP) and local legislation

Exclusion Criteria:

persistence of toxicities of prior anti cancer therapies which are deemed to be clinically relevant, known secondary malignancy requiring therapy, brain metastases which are symptomatic or require therapy, absolute neutrophil count less than 1,500/mm3, platelet count less than 100,000/mm3, haemoglobin less than 9 mg/dl, aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal, or AST or ALT greater than 5 times the upper limit of normal in case of known liver metastases, bilirubin greater than 1.5 mg/dl, serum creatinine greater than 2.0 mg/dl, concomitant intercurrent illnesses that would limit compliance with trial requirement or which are considered relevant for the evaluation of the efficacy or safety of the trial drug, chemo-, hormone- or immunotherapy within the past four weeks or within less than four half-life times of the previous drug prior to treatment with the trial drug (whatever is the longest period), radiotherapy within the past four weeks prior to treatment with the trial drug, men or women who are sexually active and unwilling to use a medically acceptable method of contraception during the trial, pregnancy or lactation, treatment with any other investigational drug within the past four weeks or within less than four half-life times of the investigational drug before treatment with the trial drug (whatever is the longest period), patient unable to comply with the protocol, patients who are considered eligible by the investigator for other second-line chemotherapy, radiotherapy or immunotherapy, patients who have received more than two lines of prior anti-tumour therapy for advanced or metastatic non small cell lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2006-07-25 (Actual); Primary Completion 2008-04-01 (Actual); Study Completion 2008-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Germany (7):
  - 1216.9.49002 Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - 1216.9.49007 Boehringer Ingelheim Investigational Site, Gauting
  - 1216.9.49008 Boehringer Ingelheim Investigational Site, Großhansdorf
  - 1216.9.49001 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1216.9.49004 Boehringer Ingelheim Investigational Site, Mainz
  - 1216.9.49005 Boehringer Ingelheim Investigational Site, Mainz
  - 1216.9.49003 Boehringer Ingelheim Investigational Site, Wiesbaden

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open-label, randomized, parallel-group, phase II clinical trial to investigate the efficacy, safety and pharmacokinetics of a single dose of 200 milligram (mg) BI 2536 administered intravenously in comparison to 50 / 60 mg BI 2536 administered intravenously on days 1, 2 and 3 in patients with advanced or metastatic non small cell lung cancer.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
  Abbreviation: Common Terminology Criteria for Adverse Events version 3.0 (CTCAE)
Groups:
- 200 Milligram (mg) BI 2536 (Day 1): A single dose of 200 mg BI 2536 on day one of each treatment course (comprising 21 days including the day of administration) was administered as an intravenous infusion over a period of 60 minutes. Each participant was planned to receive at least 2 treatment courses, in case of clinical benefit (i.e., at least stable disease and acceptable tolerability) the participants could continue therapy. Trial drug administration was stopped temporarily in case of dose limiting toxicity (DLT). Participants could continue therapy only if recovery from DLT occurred and only with a dose reduced by up to 50 mg. Dose reduction was allowed only once for a participant during the whole trial. If a participant had experienced a second episode of DLT with the reduced dose or had not recovered from DLT then the participant was withdrawn from the trial. A participant who continued therapy with BI 2536 beyond course 2 could be treated with a higher dose in case of non-progression and good tolerability.
- 50 Milligram BI 2536 (Day 1 - Day 3): A single dose of 50 mg BI 2536 on days 1, 2 and 3 of each treatment course (comprising 21 days including the days of administration) was administered as an intravenous infusion over a period of 60 minutes. Each participant was planned to receive at least 2 treatment courses, in case of clinical benefit (i.e., at least stable disease and acceptable tolerability) the participants could continue therapy with the trial drug. Trial drug administration was stopped temporarily in case of dose limiting toxicity (DLT). Participants could continue therapy only if recovery from DLT (to CTCAE levels which allowed further therapy) occurred and only with a dose reduced by up to 10 mg. Dose reduction was allowed only once for a participant during the whole trial. If a participant had experienced a second episode of DLT with the reduced dose or the participant had not recovered from DLT then the participant was withdrawn from the trial. A participant who continued therapy with BI 2536 beyond course 2 could be treated with a higher dose in case of non-progression and good tolerability.
- 60 Milligram BI 2536 (Day 1 - Day 3): After implementation of protocol amendment 2 a single dose of 60 mg BI 2536 on days 1, 2 and 3 of each treatment course (comprising 21 days including the days of administration) was administered as an intravenous infusion over a period of 60 minutes. Each participant was planned to receive at least 2 treatment courses, in case of clinical benefit (i.e., at least stable disease and acceptable tolerability) the participants could continue therapy with the trial drug. Trial drug administration was stopped temporarily in case of dose limiting toxicity (DLT). Participants could continue therapy only if recovery from DLT (to CTCAE levels which allowed further therapy) occurred and only with a dose reduced by up to 10 mg. Dose reduction was allowed only once for a participant during the whole trial. If a participant had experienced a second episode of DLT with the reduced dose or the participant had not recovered from DLT then the participant was withdrawn from the trial. A participant who continued therapy with BI 2536 beyond course 2 could be treated with a higher dose in case of non-progression and good tolerability.
Period: Overall Study
Arm/Group | 200 Milligram (mg) BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3)
Started (Entered) | 49 | 26 | 21
Treated With BI 2536 | 48 | 26 | 21
Completed | 0 | 0 | 0
Not Completed | 49 | 26 | 21
Not completed — Progressive disease | 35 | 22 | 17
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Adverse Event other than Dose Limiting Toxicity | 6 | 1 | 2
Not completed — Not treated with BI 2536 | 1 | 0 | 0
Not completed — Investigator's and participant's decision to stop treatment with BI 2536 after 6 cycles | 1 | 0 | 0
Not completed — Investigator's and participant's decision to stop treatment with BI 2536 | 1 | 0 | 0
Not completed — Investigator's decision to stop treatment with BI 2536 after 6 cycles | 2 | 0 | 0
Not completed — Investigator's decision to stop treatment with BI 2536 | 0 | 1 | 0
Not completed — Participant's decision to stop treatment with BI 2536 after 6 cycles | 0 | 0 | 1
Not completed — Participant's decision to stop treatment with BI 2536 | 2 | 0 | 1
Not completed — Increase of tumour markers | 0 | 1 | 0
Not completed — Bone metastasis | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Treated Set comprised all participants who received at least one application of the BI drug BI 2536 including treated patients who were not randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 Milligram (mg) BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Total
Number analyzed (Participants) | 48 | 26 | 21 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.8 (9.1) | 61.2 (9.1) | 62.5 (12.0) | 61.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 9 | 4 | 28
  Male | 33 | 17 | 17 | 67
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 48 | 25 | 21 | 94
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Tumour Response Evaluated According to the Response Evaluation Criteria in Solid Tumours (RECIST 1.0) by Central Review of the Tumour Images
Description: The best overall response was the best response recorded from start of treatment until the participant progressed, received any other anti-tumour therapy, died or until the individual participant's end of trial. Number of participants with 'Objective tumour response evaluated according to RECIST 1.0 by central review of the tumour images = Yes' are reported. Objective response is complete response (disappearance of all target lesions) or partial response (at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter). Changes in tumour measurements were confirmed by repeat assessments that had to be performed 6 weeks after the criteria for response had been first met.
Time Frame: assessed at baseline, then every 6 weeks (every second treatment course) until disease progression or start of any other anti-tumour therapy or death or individual participant's end of trial, up to 533 days
Population: The Treated Set comprised all participants who received at least one application of the BI drug BI 2536 including treated participants who were not randomized.
Measure: Number; unit: Number of Participants
Groups:
- Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)": A single dose of 50 mg or 60 mg (following implementation of protocol amendment 2) on days 1, 2 and 3 of each treatment course (comprising 21 days including the days of administration) was administered as an intravenous infusion over a period of 60 minutes. Each participant was planned to receive at least 2 treatment courses, in case of clinical benefit (i.e., at least stable disease and acceptable tolerability) the participants could continue therapy with the trial drug. Trial drug administration was stopped temporarily in case of dose limiting toxicity (DLT). Participants could continue therapy only if recovery from DLT (to CTCAE levels which allowed further therapy) occurred and only with a dose reduced by up to 10 mg. Dose reduction was allowed only once for a participant during the whole trial. If a participant had experienced a second episode of DLT with the reduced dose or the participant had not recovered from DLT then the participant was withdrawn from the trial. A participant who continued therapy with BI 2536 beyond course 2 could be treated with a higher dose in case of non-progression and good tolerability.
Arm/Group | 200 Milligram (mg) BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"
Number analyzed (Participants) | 48 | 26 | 21 | 47
Number of Participants | 2 | 0 | 0 | 0
Statistical Analysis 1: Comparison: 200 Milligram (mg) BI 2536 (Day 1) vs Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"; Efficacy of BI 2536 was evaluated by comparing the tumour response rate of the present trial with the tumour response rate published for patients with the same stage of disease treated with placebo. For this, treatment groups 'BI 2536 200 mg' and 'combination of treatment group 50 mg BI 2536 (day 1 - day 3) and 60 mg BI 2536 (day 1 - day 3)' were pooled together and compared to historical placebo; Test type: Other — A one-sided exact binomial test with a 2.5 % significance level was used to detect the difference between BI 2536 and historical placebo with objective response rate = 0.9 % (two out of 211) with a 95 % confidence interval of 0.2 % to 3 %; p = 0.0548, One-sided exact binomial test; Null hypothesis H0: p <= 0.009 Alternative hypothesis HA: p > 0.009

2. Secondary Outcome: Progression Free Survival
Description: Progression-free survival defined as time from date of randomisation until "date of imaging indicating progressive disease (PD) as assessed by the independent central imaging review (according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.0)" or "date of investigator assessment of clinical progression" or "date of progressive disease recorded during the follow-up period" or "death date", whatever comes first. Participants without documented progression at the time of analysis were censored at the date of the last visit.
  Per RECIST version 1.0 for target lesions and assessed by Computed Tomography (CT)-scan or Magnetic Resonance Imaging (MRI): PD, At least a 20% increase in the sum of the longest diameter (SoD) of target lesions taking as reference the smallest SoD of target lesions recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: every 6 weeks (every second treatment course), up to 419 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Groups:
- 200 Milligram BI 2536 (Day 1): A single dose of 200 mg BI 2536 on day one of each treatment course (comprising 21 days including the day of administration) was administered as an intravenous infusion over a period of 60 minutes. Each participant was planned to receive at least 2 treatment courses, in case of clinical benefit (i.e., at least stable disease and acceptable tolerability) the participants could continue therapy with the trial drug. Trial drug administration was stopped temporarily in case of dose limiting toxicity (DLT). Participants could continue therapy only if recovery from DLT (to CTCAE levels which allowed further therapy) occurred and only with a dose reduced by up to 50 mg. Dose reduction was allowed only once for a participant during the whole trial. If a participant had experienced a second episode of DLT with the reduced dose or the participant had not recovered from DLT then the participant was withdrawn from the trial. A participant who continued therapy with BI 2536 beyond course 2 could be treated with a higher dose in case of non-progression and good tolerability.
- Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3): A single dose of 50 mg or 60 mg (following implementation of protocol amendment 2) on days 1, 2 and 3 of each treatment course (comprising 21 days including the days of administration) was administered as an intravenous infusion over a period of 60 minutes. Each participant was planned to receive at least 2 treatment courses, in case of clinical benefit (i.e., at least stable disease and acceptable tolerability) the participants could continue therapy with the trial drug. Trial drug administration was stopped temporarily in case of dose limiting toxicity (DLT). Participants could continue therapy only if recovery from DLT (to CTCAE levels which allowed further therapy) occurred and only with a dose reduced by up to 10 mg. Dose reduction was allowed only once for a participant during the whole trial. If a participant had experienced a second episode of DLT with the reduced dose or the participant had not recovered from DLT then the participant was withdrawn from the trial. A participant who continued therapy with BI 2536 beyond course 2 could be treated with a higher dose in case of non-progression and good tolerability.
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 48 | 26 | 21 | 47
days | 49 [44 to 85] | 51.5 [43 to 90] | 48 [43 to 95] | 49 [44 to 85]
Statistical Analysis 1: Comparison: 200 Milligram BI 2536 (Day 1) vs Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3); Exploratory analysis. No formal hypotheses were tested; Test type: Other; p = 0.92, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.67 to 1.55] — Hazard ratio calculated as "Combination of 50 mg BI 2536 and 60 mg BI 2536" divided by 200 mg BI 2536

3. Secondary Outcome: Overall Survival
Description: Overall survival defined as time from date of randomisation until date of death from any cause. Participants alive at the time of analysis were censored at the date of the last trial visit or last date of follow-up, whatever came last.
Time Frame: every 6 weeks (every second treatment course), up to 599 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 48 | 26 | 21 | 47
days | 237 [179 to 370] | 244 [189 to 391] | 179 [102 to 244] | 196 [176 to 275]
Statistical Analysis 1: Comparison: 200 Milligram BI 2536 (Day 1) vs Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3); Exploratory analysis. No formal hypotheses were tested; Test type: Other; p = 0.65, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.7 to 1.78] — Hazard ratio calculated as "Combination of 50 mg BI 2536 and 60 mg BI 2536" divided by 200 mg BI 2536

4. Secondary Outcome: Duration of Overall Response
Description: For participants who showed an overall tumour response of complete response (CR, disappearance of all target lesions) or partial response (PR, at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter), 'duration of overall response' was defined as the time from the first date where measurement criteria were met for CR or PR (whichever was first recorded) until the first date that recurrent or progressive disease (PD) was objectively documented (taking as reference for PD the smallest measurements recorded since the treatment started). Tumour response was evaluated based on local radiological images according to RECIST version 1.0 (agreed upon by independent review). The number of participants with an CR or PR who experienced the event 'recurrent or PD' is reported instead of the time-to-event data with unit of time as the number analyzed was too small to perform a Kaplan-Meier analysis.
Time Frame: as for outcome 1
Population: All participants who received at least one application of the BI drug BI 2536 (including treated participants who were not randomized) and who showed an 'overall tumour response of complete response or partial response'.
Measure: Count of Participants; unit: Participants
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 2 | 0 | 0 | 0
Participants | 2 |  |  | 0

5. Secondary Outcome: Objective Tumour Response Evaluated According to the Response Evaluation Criteria in Solid Tumours (RECIST 1.0) by Investigator
Description: The best overall response was the best response recorded from start of treatment until the participant progressed, received any other anti-tumour therapy, died or until the individual participant's end of trial. 'Objective tumour response evaluated according to RECIST 1.0 by investigator' is 'Yes' if the best overall response is either complete response (CR, disappearance of all target lesions) or partial response (PR, at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter). Otherwise it is 'No'. To be assigned a status of 'partial response' or 'complete response', changes in tumour measurements were confirmed by repeat assessments that had to be performed six weeks after the criteria for response had been first met.
  Number of participants with 'Objective tumour response evaluated according to RECIST 1.0 by investigator = Yes' are reported.
Time Frame: as for outcome 1
Population: All participants who received at least one application of the BI drug BI 2536 (including treated participants who were not randomized) and had at least one post-baseline response evaluation.
Measure: Number; unit: Number of Participants
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"
Number analyzed (Participants) | 47 | 26 | 21 | 47
Number of Participants | 3 | 1 | 0 | 1

6. Secondary Outcome: Time-to-deterioration for Symptom Score 'Cough' Assessed on Question 1 on the Lung Cancer Module QLQ LC13 of the European Organization for Research and Treatment Quality of Life (QoL) Questionnaire (EORTC QLQ) C30 Version 3.0
Description: Time to deterioration for cough [days] was defined as the time from randomization to deterioration in score for the symptom 'cough'. Participants were considered to have deteriorated if a 10-point increase from the baseline score at any time point after baseline was observed. Participants who died before deteriorating were analyzed as having deteriorated at the time of death. Participants with disease progression without deterioration in score were censored at the time of the last scale measurement. Participants with no QoL assessments were censored at day 1. The score for symptom 'cough' was based on Question 1 on the lung cancer module QLQ LC13 of the EORTC QLQ C30 Version 3.0. A linear transformation was used to standardize the raw scores, so that scores range from 0 to 100. A high score represents a higher ("worse") level of the symptom 'cough'.
Time Frame: baseline and every 3 weeks (prior to the first administration of BI 2536 in a treatment course comprising 3 weeks), up to 539 days
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 48 | 26 | 21 | 47
days | 108 [63 to 201] | 127 [58 to 189] | 99 [74 to 179] | 102 [74 to 176]
Statistical Analysis 1: Comparison: 200 Milligram BI 2536 (Day 1) vs Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3); Test type: Other — Exploratory analysis. No formal hypotheses were tested; Regression, Cox; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.94 to 2.51] — Hazard ratio calculated as "Combination of 50 mg BI 2536 and 60 mg BI 2536" divided by 200 mg BI 2536

7. Secondary Outcome: Time-to-deterioration for Symptom Score 'Dyspnoea' Assessed on the Composite of Questions 3-5 on the Lung Cancer Module QLQ LC13 of the European Organization for Research and Treatment Quality of Life (QoL) Questionnaire (EORTC QLQ) C30 Version 3.0
Description: Time to deterioration for dyspnoea [days] was defined as the time from randomization to deterioration in score for the symptom 'dyspnoea'. Participants were considered to have deteriorated if a 10-point increase from the baseline score at any time point after baseline was observed. Participants who died before deteriorating were analyzed as having deteriorated at the time of death. Participants with disease progression without deterioration in score were censored at the time of the last scale measurement. Participants with no QoL assessments were censored at day 1. The score for symptom 'dyspnoea' was based on the composite of Questions 3-5 on the lung cancer module QLQ LC13 of the EORTC QLQ C30 Version 3.0. A linear transformation was used to standardize the raw scores, so that scores range from 0 to 100. A high score represents a higher ("worse") level of the symptom 'dyspnoea'.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 48 | 26 | 21 | 47
days | 56 [32 to 89] | 176 [93 to 198] | 80 [32 to 118] | 118 [76 to 180]
Statistical Analysis 1: Comparison: 200 Milligram BI 2536 (Day 1) vs Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3); Test type: Other — Exploratory analysis. No formal hypotheses were tested; Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.59 to 1.49] — Hazard ratio calculated as "Combination of 50 mg BI 2536 and 60 mg BI 2536" divided by 200 mg BI 2536

8. Secondary Outcome: Time-to-deterioration for Symptom Score 'Pain' Assessed on the Composite of Questions 9 and 19 of the European Organization for Research and Treatment Quality of Life (QoL) Questionnaire (EORTC QLQ) C30 Version 3.0
Description: Time to deterioration for pain [days] was defined as the time from randomization to deterioration in score for the symptom 'pain'. Participants were considered to have deteriorated if a 10-point increase from the baseline score at any time point after baseline was observed. Participants who died before deteriorating were analyzed as having deteriorated at the time of death. Participants with disease progression without deterioration in score were censored at the time of the last scale measurement. Participants with no QoL assessments will be censored at day 1. The score for symptom 'pain' was based on the composite of Questions 9 and 19 of the EORTC QLQ C30 Version 3.0. A linear transformation was used to standardize the raw scores, so that scores range from 0 to 100. A high score represents a higher ("worse") level of the symptom 'pain'.
Time Frame: as for outcome 6
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 48 | 26 | 21 | 47
days | 63 [32 to 108] | 93 [49 to 198] | 43 [22 to 102] | 76 [32 to 179]
Statistical Analysis 1: Comparison: 200 Milligram BI 2536 (Day 1) vs Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3); Test type: Other — Exploratory analysis. No formal hypotheses were tested; Regression, Cox; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.81 to 2.01] — Hazard ratio calculated as "Combination of 50 mg BI 2536 and 60 mg BI 2536" divided by 200 mg BI 2536

9. Secondary Outcome: BI 2536 Plasma Concentrations After Intravenous Infusion of 200 Milligram BI 2536 on Day 1 in Treatment Course 1
Description: BI 2536 plasma concentrations after intravenous infusion of 200 milligram BI 2536 on day 1 in treatment course 1. Geometric Coefficient of Variation reported in percentage [%].
Time Frame: on day 1 in treatment course 1: 0.5 hour (h) , 1 h, 2 h, 4 h, 120 h post-dose (planned times)
Population: The Treated Set comprised all participants who received at least one application of the BI drug BI 2536 including treated participants that were not randomized.
  Plasma concentrations below the limit of quantification were not used.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram / milliliter (ng/mL)
Arm/Group | 200 Milligram BI 2536 (Day 1)
Number analyzed (Participants) | 48
nanogram / milliliter (ng/mL)
  0.5 hour post-dose (planned time): number analyzed (Participants) | 46
  0.5 hour post-dose (planned time) | 614 (40.2)
  1 hour post-dose (planned time): number analyzed (Participants) | 47
  1 hour post-dose (planned time) | 589 (52.8)
  2 hour post-dose (planned time) | 160 (37.1)
  4 hour post-dose (planned time): number analyzed (Participants) | 47
  4 hour post-dose (planned time) | 110 (37.1)
  120 hour post-dose (planned time) | 3.07 (65.5)

10. Secondary Outcome: BI 2536 Plasma Concentrations After Intravenous Infusion of 50 / 60 Milligram BI 2536 on Day 1 in Treatment Course 1
Description: BI 2536 plasma concentrations after intravenous infusion of 50 / 60 milligram BI 2536 on day 1 in treatment course 1. Geometric Coefficient of Variation reported in percentage [%].
Time Frame: on day 1 in treatment course 1: 1 hour (h), 2 h, 23.92 h, 25 h, 47.92 h, 48.5 h, 49 h, 50 h, 52 h, 120 h post-dose (planned times)
Population: The Treated Set comprised all participants who received at least one application of the BI drug BI 2536 including treated participants who were not randomized.
  Plasma concentrations below the limit of quantification were not used.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram / milliliter (ng/mL)
Arm/Group | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 26 | 21
nanogram / milliliter (ng/mL)
  1 hour post-dose (planned time) | 114 (38.7) | 139 (70.6)
  2 hour post-dose (planned time) | 35.9 (54.6) | 39.8 (56.7)
  23.92 hour post-dose (planned time): number analyzed (Participants) | 26 | 19
  23.92 hour post-dose (planned time) | 4.89 (36.6) | 5.88 (49.5)
  25 hour post-dose (planned time): number analyzed (Participants) | 26 | 20
  25 hour post-dose (planned time) | 122 (49.4) | 152 (76.3)
  47.92 hour post-dose (planned time) | 7.21 (37.6) | 10.2 (82.4)
  48.5 hour post-dose (planned time): number analyzed (Participants) | 25 | 18
  48.5 hour post-dose (planned time) | 134 (32.4) | 170 (33.5)
  49 hour post-dose (planned time): number analyzed (Participants) | 25 | 20
  49 hour post-dose (planned time) | 121 (61.1) | 172 (63.8)
  50 hour post-dose (planned time): number analyzed (Participants) | 26 | 19
  50 hour post-dose (planned time) | 41.4 (34.6) | 51.2 (59.3)
  52 hour post-dose (planned time): number analyzed (Participants) | 26 | 20
  52 hour post-dose (planned time) | 29.2 (30.7) | 41.2 (92.0)
  120 hour post-dose (planned time): number analyzed (Participants) | 25 | 20
  120 hour post-dose (planned time) | 2.42 (53.6) | 3.19 (57.7)

11. Secondary Outcome: Incidence of Adverse Events Categorized by Common Terminology Criteria for Adverse Events (CTCAE) Grades
Description: Number of participants with adverse events categorized by "common terminology criteria for adverse events (CTCAE) grades (version 3.0)" are reported.
Time Frame: On-treatment period, that is, from first administration of the trial drug until 3 weeks after the last administration of the trial drug, up to 428 days
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 48 | 26 | 21 | 47
Participants
  Grade 1 | 7 | 6 | 2 | 8
  Grade 2 | 6 | 7 | 2 | 9
  Grade 3 | 13 | 8 | 7 | 15
  Grade 4 | 14 | 4 | 6 | 10
  Grade 5 | 6 | 1 | 4 | 5

12. Secondary Outcome: Incidence of Dose Limiting Toxicity (DLT)
Description: Dose limiting toxicity was defined as drug related common terminology criteria for adverse events (CTCAE) grade 3 or greater non haematological toxicity (excluding untreated nausea, vomiting or diarrhoea) or drug related CTCAE grade 4 neutropenia for seven or more days and / or complicated by infection or CTCAE grade 4 thrombocytopenia. Number of participants with DLT is reported.
Time Frame: as for outcome 11
Population: as for outcome 1
Measure: Number; unit: Participant
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of 50 mg BI 2536 (Day 1 - Day 3) and 60 mg BI 2536 (Day 1 - Day 3)
Number analyzed (Participants) | 48 | 26 | 21 | 47
Participant | 8 | 4 | 3 | 7

13. Secondary Outcome: Number of Participants With Neutropenia of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4
Description: Number of participants with neutropenia of common terminology criteria for adverse events (CTCAE) grade 3 or 4.
Time Frame: as for outcome 11
Population: The Treated Set comprised all participants who received at least one application of the BI drug BI 2536 including treated participants who were not randomized.
  Participants with laboratory values that were out of range for CTCAE grading and were deemed possible clinically significant abnormal were excluded from the analyses.
Measure: Number; unit: Number of Participants
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"
Number analyzed (Participants) | 46 | 26 | 20 | 46
Number of Participants | 33 | 6 | 12 | 18

14. Secondary Outcome: Number of Participants With Thrombocytopenia of Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or 4
Description: Number of participants with thrombocytopenia of common terminology criteria for adverse events (CTCAE) grade 3 or 4.
Time Frame: as for outcome 11
Population: as for outcome 13
Measure: Number; unit: Number of Participants
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"
Number analyzed (Participants) | 42 | 24 | 20 | 44
Number of Participants | 4 | 1 | 0 | 1

15. Secondary Outcome: Change From Baseline in Systolic/Diastolic Blood Pressure at Individual Participant's End-of-trial Visit
Description: Change from baseline in systolic/diastolic blood pressure at individual participant's end-of-trial visit.
Time Frame: baseline, date of individual participant's end of trial visit which was 533 days after start of treatment at the latest
Population: All participants who received at least one application of the BI drug BI 2536 (including treated patients who were not randomized) and for whom data were collected for this endpoint at the end-of-trial visit.
Measure: Mean (Standard Deviation); unit: millimetre of mercury (mmHg)
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"
Number analyzed (Participants) | 15 | 14 | 7 | 21
millimetre of mercury (mmHg)
  Change from baseline in systolic blood pressure | 2.4 (16.6) | -2.4 (14.0) | 2.9 (17.8) | -0.7 (15.1)
  Change from baseline in diastolic blood pressure | -2.0 (14.7) | 0.8 (13.7) | -7.1 (12.5) | -1.9 (13.5)

16. Secondary Outcome: Change From Baseline in Pulse Rate at Individual Participant's End-of-trial Visit
Description: Change from baseline in pulse rate at individual participant's end-of-trial visit.
Time Frame: baseline, date of individual participant's end of trial visit which was 533 days after start of treatment at the latest
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | 200 Milligram BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"
Number analyzed (Participants) | 14 | 13 | 6 | 19
beats per minute (bpm) | 10.6 (14.3) | 4.5 (13.3) | -8.0 (14.1) | 0.5 (14.4)

ADVERSE EVENTS:
Time Frame: For Serious and Other Adverse Events: On-treatment period, that is, from first administration of the trial drug until 3 weeks after the last administration of the trial drug, up to 428 days. For All-Cause Mortality: On-treatment period + Follow-up period, up to 599 days.
Description: All participants who received at least one dose of BI 2536 were included in the safety analyses.
Groups:
- 200 Milligram (mg) BI 2536 (Day 1): A single dose of 200 mg BI 2536 on day one of each treatment course (comprising 21 days including the day of administration) was administered as an intravenous infusion over a period of 60 minutes. Each participant was planned to receive at least 2 treatment courses, in case of clinical benefit (i.e., at least stable disease and acceptable tolerability) the participants could continue therapy with the trial drug. Trial drug administration was stopped temporarily in case of dose limiting toxicity (DLT). Participants could continue therapy only if recovery from DLT (to CTCAE levels which allowed further therapy) occurred and only with a dose reduced by up to 50 mg. Dose reduction was allowed only once for a participant during the whole trial. If a participant had experienced a second episode of DLT with the reduced dose or the participant had not recovered from DLT then the participant was withdrawn from the trial. A participant who continued therapy with BI 2536 beyond course 2 could be treated with a higher dose in case of non-progression and good tolerability.
Arm/Group | 200 Milligram (mg) BI 2536 (Day 1) | 50 Milligram BI 2536 (Day 1 - Day 3) | 60 Milligram BI 2536 (Day 1 - Day 3) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)"
All-Cause Mortality (participants affected / at risk) | 35/48 | 20/26 | 16/21 | 36/47
Serious Adverse Events (participants affected / at risk) | 20/48 | 8/26 | 12/21 | 20/47
Other Adverse Events (participants affected / at risk) | 44/48 | 24/26 | 19/21 | 43/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 200 Milligram (mg) BI 2536 (Day 1) (N=48) | 50 Milligram BI 2536 (Day 1 - Day 3) (N=26) | 60 Milligram BI 2536 (Day 1 - Day 3) (N=21) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)" (N=47)
Anaemia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1
Right ventricular failure (Cardiac disorders) | 1 | 0 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 1
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 3 | 2 | 5
Respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Catheter removal (Surgical and medical procedures) | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 200 Milligram (mg) BI 2536 (Day 1) (N=48) | 50 Milligram BI 2536 (Day 1 - Day 3) (N=26) | 60 Milligram BI 2536 (Day 1 - Day 3) (N=21) | Combination of Treatment Group "50 mg BI 2536 (Day 1 - Day 3)" and "60 mg BI 2536 (Day 1 - Day 3)" (N=47)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 3
Leukopenia (Blood and lymphatic system disorders) | 4 | 0 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 16 | 2 | 5 | 7
Vertigo (Ear and labyrinth disorders) | 5 | 4 | 1 | 5
Constipation (Gastrointestinal disorders) | 10 | 5 | 4 | 9
Diarrhoea (Gastrointestinal disorders) | 7 | 5 | 3 | 8
Nausea (Gastrointestinal disorders) | 15 | 6 | 4 | 10
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 9 | 0 | 3 | 3
Asthenia (General disorders) | 4 | 1 | 1 | 2
Chest pain (General disorders) | 6 | 2 | 0 | 2
Chills (General disorders) | 0 | 1 | 2 | 3
Fatigue (General disorders) | 14 | 10 | 5 | 15
Injection site phlebitis (General disorders) | 0 | 2 | 0 | 2
Injection site reaction (General disorders) | 0 | 3 | 2 | 5
Oedema (General disorders) | 0 | 0 | 2 | 2
Oedema peripheral (General disorders) | 6 | 1 | 3 | 4
Pyrexia (General disorders) | 3 | 1 | 2 | 3
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 2
Nasopharyngitis (Infections and infestations) | 8 | 6 | 0 | 6
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 4
C-reactive protein increased (Investigations) | 3 | 0 | 1 | 1
Weight decreased (Investigations) | 3 | 1 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 9 | 2 | 4 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1 | 2
Headache (Nervous system disorders) | 7 | 3 | 2 | 5
Paraesthesia (Nervous system disorders) | 0 | 2 | 0 | 2
Polyneuropathy (Nervous system disorders) | 3 | 2 | 2 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 6 | 2 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 2 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 0 | 4 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 1 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 4 | 2 | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 3
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Phlebitis (Vascular disorders) | 1 | 2 | 2 | 4
Thrombophlebitis (Vascular disorders) | 1 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.